CLINICAL TRIAL: NCT03549936
Title: Role of Low Lactose Infant Formula In The Management of Neonatal Abstinence Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Dr Deepak Kumar, Neonatologist, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB14-00005
Record Dates: First submitted 2017-05-06; First posted 2018-06-08 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: NAS, low lactose formula
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind Clinical trial on Role of Low Lactose Formula In the Management of Neonatal Abstinence Syndrome
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Infants who develop NAS will continue to receive blinded formula as part of non-pharmacological treatment and will also receive pharmacological treatment (morphine/methadone) as per hospital guidelines directed by their medical care providers. Pharmacological treatment will be optimized and weaned as per standard hospital guidelines. Use of blinded formula A or B will be continued until 2 weeks of age at which point its use as study intervention will be completed. After this point, parents/home care providers and medical care providers may use formula of their preference. However we will offer them a choice of continuing the blinded formula until the infant is discharged at which point standard formula will have to be initiated. General clinical data will be collected at discharge including length of stay and weight.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low lactose formula (Active Comparator): If infant is not breast feeding and parents plan to formula feed, following written informed consent, infant is randomized to receive "low lactose formula" which arrives from milk lab labeled as formula "A" or formula "B".
  Interventions: Other: Low lactose or regular formula
- Regular formula (Active Comparator): If infant is not breast feeding and parents plan to formula feed, following written informed consent, infant is randomized to receive "regular formula" which arrives from milk lab labeled as formula "A" or formula "B"
  Interventions: Other: Low lactose or regular formula

INTERVENTIONS:
Other: Low lactose or regular formula — If infant is not breast feeding and parents plan to formula feed, following written informed consent, infant is randomized to receive "low lactose formula" or "regular formula" which arrives from milk lab blinded and labeled as formula "A" or formula "B".

SUMMARY:
Currently Morphine and or Methadone are the most commonly used drugs in the treatment for NAS along with supportive care. Many care providers offer tolerance "low lactose" formula to these infants to alleviate gastrointestinal symptoms. There are no clinical studies to support this practice and it is currently unknown that low lactose formula really helps or not in management of NAS.

This is a Randomized Double Blind Clinical Trial to assess the role of low lactose formula versus standard (regular) formula in managing NAS.

DETAILED DESCRIPTION:
At birth, and after written informed consent, investigators will encourage opiate dependent mothers to breast feed if appropriate in accordance with hospital NAS management guidelines (sober for at least 4-6 months, enrolled in a drug treatment program, HIV negative). If mother is unable to breast feed and or chooses formula feeding for the infant or the infant needs supplemental formula due to inadequate lactation or poor weight gain, then the infant will be randomized to either receive blinded "low lactose formula Similac Sensitive" or "regular cow mild based formula Similac Advance". These will be simply labelled as Formula A and formula B. The randomization will be done using computer generated random number coupled with stratified balanced blocked methodology. Recent reformulations by Abbott Nutrition in the US market nation wide has resulted in "low lactose formula Similac Sensitive" being made 19 cal/oz or 20 cal/oz or "regular cow mild based formula Similac Advance" which is now only available as 19 cal/oz instead of 20 cal/oz. This change in calorie density has occured to reflect newer data suggested that human breast milk has 19 cal/oz instead of 20 cal/oz as believed previously. Abbott has continued to make 20 cal/oz Similac sensitive because many many providers across the country are using this for NAS babies. There are some differences in other carbohydrates other than lactose (both have <1% lactose) in the two Similac Sensitive 19 and 20 cal/oz. The calorie difference is of no clinical significance in term infants because they modulate their volume of milk consumed.

After recruitment and randomization at birth, infants will be fed every 2-3 hrs or on demand and will also be observed for NAS score every 2-3 hours starting soon after birth. Infants will receive their "medical provider directed" standard pharmacological and non-pharmacological treatment.

Those who do not demonstrate NAS, will be discharged after 5-7 days of observation. Study formula will be discontinued or may be continued if they or their provider chose to do so.

Infants who develop NAS will continue to receive blinded formula as part of non-pharmacological treatment and will also receive pharmacological treatment (morphine/methadone) as per hospital guidelines directed by their medical care providers. Pharmacological treatment will be optimized and weaned as per standard hospital guidelines. Use of blinded formula A or B will be continued until 2 weeks of age at which point its use as study intervention will be completed. After this point, parents and medical care providers may use formula of their preference. However investigators will offer a choice of continuing the blinded formula until the infant is discharged at which point standard formula will have to be initiated. General clinical data will be collected at discharge including length of stay and weight.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine exposure of opiate and related drugs-morphine
* Late preterm or full term (36-42 weeks of gestation)

Exclusion Criteria:

* Major congenital anomalies
* Post-surgical cases
* Major respiratory, cardiovascular, neurological or metabolic disorders
* Less than 36 completed weeks of gestation

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of morphine required to treat NAS. | 14 days of age
  Every dose of morphine required to treat NAS over first 14 days of life will be noted and total cumulative dose administered will be observed. We expect infants on low lactose formula versus regular formula will require lower cumulative dose of morphine during first 2 weeks of life.
Highest dose of morphine required to treat NAS. | 14 days of age
  Every dose of morphine required to treat NAS over first 14 days of life will be noted. We expect infants on low lactose formula versus regular formula will require lower maximal dose of morphine.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kumar, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pahl A, Young L, Buus-Frank ME, Marcellus L, Soll R. Non-pharmacological care for opioid withdrawal in newborns. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD013217. doi: 10.1002/14651858.CD013217.pub2. PMID 33348423